CLINICAL TRIAL: NCT06190522
Title: Diagnosis of Acute Obstructive Renal Failure by Clinical Ultrasound Performed by the Emergency Physician.
Acronym: IRASMU
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0118; 2021-A00777-34 (Other: ID-RCB)
Record Dates: First submitted 2023-12-14; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Failure
Keywords: acute renal failure; ultrasound; diagnosis
MeSH Terms: conditions — Acute Kidney Injury; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute renal failure: Patients receiving a clinical ultrasound by the on-site emergency physician trained in the technique
  Interventions: Diagnostic Test: Emergency physician clinical ultrasound

INTERVENTIONS:
Diagnostic Test: Emergency physician clinical ultrasound — Clinical ultrasound by emergency doctor consisting in obtaining frontal sections of the 2 kidneys and a transverse section of the bladder

SUMMARY:
Acute renal failure is frequently diagnosed in the emergency room during a biological assessment. Its discovery requires determining the cause, which may be either functional, or obstructive. The obstructive cause is responsible for 10% of acute renal failure. It is recommended to start the exploration of this pathology with an ultrasound in search of an obstructive cause. However, ultrasound from the radiologist is not always available.

The realization of this ultrasound by the emergency physician would reduce the time to obtain the diagnosis and therefore the time of passage to the emergency room.

No study has yet been carried out to validate the performance of this ultrasound by the emergency physician in the case of acute renal failure.

This study would validate the diagnostic performance of this ultrasound technique in order to identify as quickly as possible patients with acute renal failure whose cause is obstructive.

DETAILED DESCRIPTION:
Acute renal failure is frequently diagnosed in the emergency room during a biological assessment. Its discovery requires determining the cause, which may be either functional, i.e. kidney dysfunction, or obstructive. The obstructive cause is responsible for 10% of acute renal failure. It is recommended to start the exploration of this pathology with an ultrasound in search of an obstructive cause. However, ultrasound from the radiologist is not always available.

The realization of this ultrasound by the emergency physician would reduce the time to obtain the diagnosis and therefore the time of passage to the emergency room.

No study has yet been carried out to validate the performance of this ultrasound by the emergency physician in the case of acute renal failure.

The aim of this research is to evaluate the performance of clinical ultrasound in the diagnosis of an obstructive cause of acute renal failure by the emergency physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an emergency structure
* Patients with acute renal failure (defined by an increase of 1.5 x the baseline serum creatinine value (known or expected according to age and sex))

Exclusion Criteria:

* Patients unable to express their non-objection
* Patients who have undergone a kidney transplant
* Dialysis patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute renal failure recruited during their visit to the emergency department where the ultrasound will be performed
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Performance of clinical ultrasound diagnosis by the emergency physician | Up to 2 weeks
  Performance (sensitivity and specificity) of the diagnosis of an obstructive cause of acute renal failure by emergency physicians performing clinical ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Frederic BALEN, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hudson KB, Sinert R. Renal failure: emergency evaluation and management. Emerg Med Clin North Am. 2011 Aug;29(3):569-85. doi: 10.1016/j.emc.2011.04.005. PMID 21782075
- [Background] Liano F, Pascual J. Epidemiology of acute renal failure: a prospective, multicenter, community-based study. Madrid Acute Renal Failure Study Group. Kidney Int. 1996 Sep;50(3):811-8. doi: 10.1038/ki.1996.380. PMID 8872955
- [Background] Pathan SA, Mitra B, Mirza S, Momin U, Ahmed Z, Andraous LG, Shukla D, Shariff MY, Makki MM, George TT, Khan SS, Thomas SH, Cameron PA. Emergency Physician Interpretation of Point-of-care Ultrasound for Identifying and Grading of Hydronephrosis in Renal Colic Compared With Consensus Interpretation by Emergency Radiologists. Acad Emerg Med. 2018 Oct;25(10):1129-1137. doi: 10.1111/acem.13432. Epub 2018 May 28. PMID 29663580
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Derived] Balen F, Drumare L, Laclergerie F, Gaudreau-Simard M, Guy P, Dubucs X. Diagnostic accuracy of point-of-care ultrasonography for obstructive cause in patients with acute kidney injury: a prospective diagnosis cohort. Intern Emerg Med. 2025 Jun 8. doi: 10.1007/s11739-025-03996-2. Online ahead of print. PMID 40483617